CLINICAL TRIAL: NCT03698396
Title: A Phase I/II, Open-Arm Study Evaluating the Safety of Islet Transplant in Patients With Type I Diabetes
Brief Title: Islet Transplant in Patients With Type I Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kenneth Brayman, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Brayman, MD, Professor, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170020
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogenic Islet Cell Transplantation (Experimental): Transplantation of allogenic islet cell will be given to eligible patients, up to three times during the study, using cell quantities based on body weight.
  Interventions: Biological: Allogenic Islet Cell Transplantation

INTERVENTIONS:
Biological: Allogenic Islet Cell Transplantation — Transplantation of allogenic islet cells will be given to eligible patients, up to three times during the study, using cell quantities based on body weight.

SUMMARY:
The primary objective of this study is to demonstrate the safety of allogenic islet transplantation in type 1 diabetic patients performed at the University of Virginia.

The purpose is to demonstrate that islet transplantation can be performed safely and reliably achieves better glycemic control than state-of-the-art insulin treatment in management of type 1 diabetic patients with brittle control and a history of severe hypoglycemic episodes with hypoglycemia unawareness.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is caused by islet autoimmunity followed by immune destruction of the β-cells. In 2015 the International Diabetes Federation reported that 36 million people suffer from T1D globally, while it is estimated that 1.4 millions of Americans have T1D. Although life expectancy of patients with T1D has much improved since the introduction of insulin therapy, chronic complications, including blindness and renal failure, are hampering the quality of life and represent a multi-billion dollar annual burden on the health care system of industrialized countries. Keeping blood glucose levels under tight control represents the most effective way either to prevent the onset or to reduce the progression of the chronic complications of T1D. At present, such a goal may be accomplished by treating patients with intensified therapy regimens consisting of multiple insulin injections, which involve accurate blood glucose monitoring. However, administration of subcutaneous insulin can never approximate pulsatile insulin secretory patterns of the normal β-cells, and rarely attains normal blood glucose levels without the risk of major hypoglycemic episodes. In addition, intensive insulin therapy is only suitable for selected patients.

Pancreas transplantation is an alternative therapeutic modality which can stop the progression of diabetic complications without increasing the incidence of hypoglycemic events. Unfortunately, this procedure, usually performed simultaneously with a kidney graft, has a high morbidity and a significant mortality rate. Pancreas transplantation, in spite of an important impact on the quality of life in successful cases, is often restricted to selected patients. In this context, islet transplantation offers and alternative treatment solution, normalizing glucose metabolism without the risk of hypoglycemia and avoiding the potentially life threatening complications of whole pancreas grafts.

Clinical islet transplantation has continuously advanced over the past two decades, with clear improvements in islet manufacturing and clinical outcomes, therefore restore insulin production and ameliorate glycemic instability in patients with T1D. Currently, the procedure is primarily indicated for patients with a history of life threatening severe hypoglycemia and hypoglycemia unawareness for which islet transplantation has been highly effective both in the short and long terms. According to the most recent public presentation from the collaborative islet transplant registry (CITR), 1055 allogeneic islet transplantations have been reported by 50 islet transplantation centers in North America, Europe, Australia, and South Korea. Of these cases, islet transplant alone was the most frequent procedure (n=858) followed by islet after kidney (IAK) and simultaneous islet and kidney transplantation (SIK) (n=197). CITR data has identified factors that predict the achievement and maintenance of insulin independence as recipient age over 35 years, more than half a million infused islet equivalent (IEQ), islet glucose stimulation index >1.5, induction therapy with Tcell depletion, and TNF-α inhibitor and maintenance with calcineurin inhibitor and mTOR inhibition. The combination of these factors in 60 recipients resulted in stable insulin independence after 5 years in 60 % of the patients. Recipient age, IEQ, and calcineurin inhibitor (CNI) maintenance were also predictive of positive C-peptide levels (≥0.3 ng/ml; n=308) and HbA1c (<6.5 % or drop ≥2 %; n=530) and age and IEQ predicted absence of severe hypoglycemic events (SHE) (>90 % of patients at 5 years). As another indicator of improvements in the procedure, the number of adverse events has dropped significantly in the past 5 years, with 80 % free of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 episode of severe hypoglycemia in the past 3 years
* Reduced awareness of hypoglycemia
* Must be a qualified candidate for pancreas transplant

Exclusion Criteria:

* Diagnosis of co-existing cardiac diseased (ie, recent myocardial infarction within 6 months or angiographic evidence of non-correctable coronary artery disease or evidence of ischemia on functional cardiac exam
* Active alcohol or substance abuse
* Psychiatric disorder this is unstable or uncontrolled on current medication
* History of non-compliance
* Active infection including hepatitis C, hepatitis B, HIV
* History of or active Tuberculosis
* Any history of cancer, except skin cancer
* History of stroke within past 6 months
* BMI > 27 kg/m2
* C-peptide fasting response to glucagon stimulation
* Inability to provide informed consent
* Creatinine Clearance < 60 ml/min
* Macroalbuminuria
* Baseline Hb <12 gm/dL
* Baseline liver function test outside normal ranges
* History of untreated proliferative retinopathy
* Positive pregnancy test or male subjects intent to procreate while on study
* Previous transplant (except islet transplant)
* Insulin requirement of > 0.7 IU/kg/day
* HbA1c . 12%
* Hyperlipidemia
* Under treatment for medical condition requiring chronic use of steroids
* Use of coumadin or other antiplatelet therapy
* History of Factor V deficiency
* History of Addison's disease
* Allergic to radiographic contrast material
* Symptomatic cholecystolithiasis
* Acute on chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Treatment with antidiabetic medication other than insulin within 4 weeks of enrollment
* Use of any investigational drug or device within 4 weeks of enrollment
* Received a live attenuated vaccine within 2 months of listing
* Active coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure related adverse events | within 1 year of transplant
  as evidenced by lack of bleeding during the procedure, incidence of portal vein thrombosis, incidence of biliary puncture during the procedure, incidence of wound complication for cases where laparotomy is performed, and incidence of increased transaminase levels >5 times upper limit of normal within 6 months.

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c less than or equal to 7.0% | within 1 year of transplant
  Measured by IV venous blood draw
Proportion of subjects free of severe hypoglycemic events between 6 and 12 months from the time of first islet cell infusion or from the time insulin therapy is withdrawn | within 1 year of transplant
  An event with symptoms compatible with hypoglycemia in which the subject required assistance of another person and which was associated with either a blood glucose level of <50 mg/dl or prompt recovery after oral carbohydrate, intravenous glucose or glucagon administration.
Insulin independence achieved | within 1 year of transplant
  Measured by absence of exogenous insulin injection, HbA1c less than or equal to 7.0%, fasting capillary glucose level that does not exceed 140 mg/dl more than three times per week during a seven day period, and fasting plasma glucose levels less than or equal to 126 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No